CLINICAL TRIAL: NCT00148720
Title: A Phase II Study of Preoperative Capecitabine in Women With Operable Breast Cancer
Brief Title: Capecitabine in Women With Operable Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Hoffmann-La Roche (Industry); Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Ian E. Krop, MD, PhD, Assistant Professor of Medicine, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-167
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Invasive Breast Carcinoma; Primary Invasive Breast Cancer; Stage I Breast Cancer; Stage II Breast Cancer; Stage III Breast Cancer
Keywords: Invasive Breast Cancer; Operable Breast Cancer; Capecitabine
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

INTERVENTIONS:
Drug: Capecitabine — Taken orally twice a day for 14 days and treatment will repeat every 21 days (1 cycle) for 4 cycles

SUMMARY:
The purpose of this study is to find out what effects (good and bad) taking capecitabine for 12 weeks before surgery will have on women with breast cancer.

DETAILED DESCRIPTION:
* Prior to the start of treatment, patients will have a small metal clip inserted into the tumor bed to identify the tumor site to the surgeon. At that time, a needle biopsy of the breast tumor or a sentinel (underarm) lymph node biopsy will also be performed.
* Patients will take capecitabine orally twice daily for 14 days. This treatment will repeat every 21 days (1 cycle). Patients will receive 4 cycles of this treatment.
* A physical exam and blood work will be done every three weeks after starting therapy to monitor side effects.
* After two weeks of capecitabine a biopsy from the tumor will be done to generate information about the characteristics of the tumor that may respond to capecitabine.
* After completing 4 cycles (12 weeks) of capecitabine, patients will then undergo surgery to remove any remaining breast cancer (lumpectomy or mastectomy). Post-surgical treatment (radiation, chemotherapy, and hormonal therapy) is at the discretion of the patients physician.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of primary invasive breast cancer
* Stage I-III operable breast cancer.
* Primary tumor must be greater than or equal to 2cm by radiographic imaging or palpitation
* Women greater than 18 years of age
* ECOG performance status 0-1
* WBC > 4000/mm3
* Platelet count > 100,000/mm3
* SGOT < 2x ULN
* Calculated creatinine clearance > 50ml/min

Exclusion Criteria:

* Evidence of metastatic (stage IV) cancer on physical exam or any diagnostic study.
* Pregnant or breast-feeding women
* Inflammatory breast cancer
* HER2 positive disease
* History of hypersensitivity to a 5-FU or known dihydropyrimidine dehydrogenase (DPD) deficiency
* Uncontrolled intercurrent illness
* Prior history of breast cancer are ineligible except: diagnosed at least 2 years ago; present cancer is not in previously irradiated breast; no prior chemotherapy in the past 5 years; no prior high-dose chemotherapy with stem cell or bone marrow transplant.
* Excisional biopsy performed prior to enrollment
* Uncontrolled coagulopathy
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2004-09; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To determine the response rate following four cycles of preoperative capecitabine in women with operable breast cancer. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ian Krop, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Faulkner Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Result] Tolaney SM, Jeong J, Guo H, Brock J, Morganstern D, Come SE, Golshan M, Bellon J, Winer EP, Krop IE. A phase II study of preoperative capecitabine in women with operable hormone receptor positive breast cancer. Cancer Med. 2014 Apr;3(2):293-9. doi: 10.1002/cam4.164. Epub 2014 Jan 27. PMID 24464780